CLINICAL TRIAL: NCT03736590
Title: The Effect of a Clinic-Based Financial Coaching on Health and Development
Brief Title: Clinic-Based Financial Coaching and Family Health and Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Adam Schickedanz, Assistant Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UCLAHarborSchickedanzMFP
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Economic Problems; Development, Child; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Pediatricians and outcomes assessors will not be aware of study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Financial Coaching Plus Social Needs Screening (Experimental): Families in this intervention arm will receive financial coaching at each well child visit, in addition to clinic-based social needs screening and referral.
  Interventions: Behavioral: Financial coaching and services
- Control - Social Needs Screening and Referral (Active Comparator): Families in this active control arm will receive social needs screening and referral to community resources to address identified social needs.
  Interventions: Behavioral: Financial coaching and services

INTERVENTIONS:
Behavioral: Financial coaching and services — The intervention will consist of clinic-based financial coaching that focuses on improving financial stability through longitudinal visits with financial services professionals to address financial goals.

SUMMARY:
This study will examine the impact of clinic-based financial coaching on parent health-related quality of life and child development measures, as well as family social needs for families with young children receiving pediatric care at a primary care practice in the Los Angeles County safety net.

DETAILED DESCRIPTION:
With an expert group of researchers, financial coaches, and implementation scientists, we will study the impact of clinic-based financial coaching on parent health-related quality of life, child developmental risk, and social needs.We will conduct a clinical randomized controlled trial of financial coaching for low-income families. Parents of infants in a large pediatric primary care safety-net clinic will receive either 1) financial coaching from trained coaches plus social needs screening and resource navigation at all well child visits (intervention) or 2) social needs screening and navigation alone (active control) and will be followed for five years. Aims include:

1a) Examine parent outcomes of overall health-related quality of life (primary parent outcome);

1b) Examine child outcomes of developmental risk scores (primary child outcome) and well-child visit adherence;

1c) Examine family social needs outcomes, including incidence of any food insecurity, housing instability, transportation or utilities interruptions (primary family outcome any one or more) and resource use; and financial metrics.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers in families with children 4 months or under at enrollment receiving care at Harbor-UCLA medical center clinic.

Exclusion Criteria:

* Cognitive impairment or not speaking English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQOL) - Patient Reported Outcome Measurement Information System Global Health Short Form 10-Item Scale (PROMIS-10) | Interval change in PROMIS-10 HRQOL will be assessed over up to a 5 year period.
  Health-related quality of life will be measured at baseline and regular intervals using the Patient-Reported Outcomes Measurement Information System Global Health Short Form 10 (PROMIS 10). This will be the primary outcome for parents in the study. The PROMIS-10 measures overall health, physical health, mental health and social functioning and is scored on a T-scored range with 50 as the mean and 10 as the standard deviation. Higher scores indicate better HRQOL.
Developmental Risk - Ages and Stages Questionnaires | Interval change in developmental risk will be assessed over up to a 5 year period.
  Parent report of child developmental risk via clinic-based developmental questionnaires (Ages and Stages Questionnaires, ASQ) will be used to measure developmental risk. The ASQ measure contains sub-scales for each developmental domain (gross motor, fine motor, problem solving, communication, problem-solving, personal-social). Parent-reported ASQ items yield a score from 0-60 with cutoffs determining children at risk for developmental delay. Higher scores indicate less risk of developmental delay.
Presence of Any Social Need - Accountable Health Communities Social Needs Screening Items | Interval change in presence of any social need will be assessed over up to a 5 year period.
  Family social needs to be assessed at baseline and regular intervals include food insecurity, housing insecurity, transportation problems, utilities problems, and legal issues. All of these social needs are measured using the Accountable Health Communities Social Needs Screener and the presence of any of the above social needs will be interpreted as the presence of a social need. Social needs resource use will also be measured.

SECONDARY OUTCOMES:
Economic Stress - Family Economic Strain Scale. | Interval change in FESS will be assessed over up to a 5 year period.
  Family economic stress will be measured using the Family Economic Strain Scale (FESS) score. The FESS has 15 items and ranges from a score of 5 to 75, with higher scores indicating less financial stress.
Parenting Self-Efficacy - Parenting Sense of Competence Scale | Interval change in PSOC will be assessed over up to a 5 year period.
  Parenting self-efficacy will be measured using the Parenting Sense of Competence Scale (PSOC). The PSOC is a 17 item scale with a range from 17 to 102, with higher scores indicating more parent competence.
Pediatric Primary Care Visit Adherence | Interval change in pediatric primary care visit adherence will be assessed over up to a 5 year period.
  Pediatric primary care visit adherence will be measured as a rate for families in the study.

OTHER OUTCOMES:
Financial Measures - Income | Interval change in financial measures will be assessed over up to a 5 year period.
  Family financial measure of dollar value of yearly income will be collected via survey.
Financial Measures - Savings | Interval change in financial measures will be assessed over up to a 5 year period.
  Family financial measure of dollar value of savings will be collected as part of the study via survey.
Financial Measures - Debt | Interval change in financial measures will be assessed over up to a 5 year period.
  Family financial measure of dollar value of debt will be collected as part of the study via survey.
Financial Measures - Credit Score | Interval change in financial measures will be assessed over up to a 5 year period.
  Family financial credit score will be collected as part of the study via survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Adam Schickedanz, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No